CLINICAL TRIAL: NCT03506594
Title: Radiofrequency Non-ablative in the Treatment of Genitourinary Syndrome of Menopause
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Centro de Atenção AP
Record Dates: First submitted 2018-03-15; First posted 2018-04-24 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Genitourinary Syndrome of Menopause

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency ON and Kinesiotherapy (Active Comparator): The radiofrequency application protocol with the CAPENERGY device, which has two electrodes: an active one, which will be introduced into the vagina, using a condom and gel to the emission of radiofrequency and another electrode, dispersive, coupled to the patient's hip, which will function as earth. The temperature used in the treatment will be 41°C, which this parameter will be placed in the equipment, maintained for 2 minutes at the anterior wall and 2 others minutes at the posterior wall. Five RF sessions will be performed, with a seven-day interval between them. For the application, participants will be placed in supine position. The session will be quick, with an average duration of 20 minutes. Kinesiotherapy will be done once a week, totaling five sessions. Initially, verbal information about location, function, and the correct way to contract the pelvic floor (PA) will be given.
  Interventions: Device: Radiofrequency non ablative
- Radiofrequency OFF and Kinesiotherapy (Placebo Comparator): The patient will be in supine decubitus, the vaginal probe of the radiofrequency apparatus will be introduced, with the gel previously heated. The radiofrequency will be off.
  Kinesiotherapy will be done once a week, totaling five sessions. Initially, verbal information about location, function, and the correct way to contract the pelvic floor (PA) will be given.
  Interventions: Device: Radiofrequency non ablative

INTERVENTIONS:
Device: Radiofrequency non ablative — The application of RF was performed by physical therapist trained in the technique of radiofrequency through the CAPENERGY device with capacitive transfer method using non-ablative handle with active electrode placed intra-vaginal and coupling electrode placed on the participant's back. For application, the participants were in gynecological position. The session had an average duration above 20 minutes. The temperature was measured by an infrared thermometer and when it reached 41°C radiofrequency was maintained for 2 minutes in the anterior wall and 2 other minutes in the posterior wall of the vagina.

SUMMARY:
The study is conducted in women at the menopause with a clinical diagnosis of Genitourinary Syndrome, which presents symptoms in of vulvovaginal atrophy and tract urinary and were treated with radiofrequency non ablative technique for capacitive transfer in intra-vaginal. All participants were evaluated by a physical therapist and did the exam of PH vaginal, cell maturation index and questionnaires. The participants made five sessions of Radio Frequency (RF) with an interval of seven days between them. The application of RF was performed by physical therapist trained in the technique of radio frequency through the Capenergie brand device with capacitive transfer method using non-ablative handle with active electrode intra-vaginal and coupling electrode placed on the participant's back. For application, the participants were in gynecological position. The session had an average duration above 20 minutes. The temperature was measured by an infrared thermometer when it reached 41graus radiofrequency was maintained for 2 minutes in the anterior wall and 2 minutes more in the posterior wall of vagina.

ELIGIBILITY:
Inclusion Criteria:

* will be women in menopause until 65 years of age with clinical complaints of Genitourinary Syndrome of Menopause and who agree to voluntarily participate in the research.

Exclusion Criteria:

* will be excluded from the study participants with limited understanding, with neurological degenerative chronic diseases, sensory deficit in the genital region, users of pacemaker and intrauterine device of cooper and women under hormone therapy under six months

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Change in Cell maturation index | Each 3 months pos treatment, until one year
  % cells parabasal, % intermediate cells and superficial cells
Change in Vaginal PH | Each 3 months pos treatment, until one year
  During the fertile years of life, the vaginal pH ranges from 3.5 to 4.5. At menopause, vaginal Ph increases to above 4.5. The higher the vaginal Ph, the greater the degree of atrophy

SECONDARY OUTCOMES:
Numeric Visual Scale | one week, one month, three months, six months, nine months and one year
  Will be evaluated vaginal dryness, pain during intercourse, vaginal laxity, burning sensation and itching, on a scale of 0 to 10, being 0 asymptomatic and 10 the maximum of symptoms
Questionnaire of quality of life specified urinary incontinence | one week, one month, three months, six months, nine months and one year
  The ICIQ-SF
Female Sexual Function Index | one week, one month, three months, six months, nine months and one year
  FSFI
Female Genital Self-image Scale | one week, one month, three months, six months, nine months and one year

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Atenção ao Assoalho Pelvico, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinheiro C, Costa T, Amorim de Jesus R, Campos R, Brim R, Teles A, Vilas Boas A, Lordelo P. Intravaginal nonablative radiofrequency in the treatment of genitourinary syndrome of menopause symptoms: a single-arm pilot study. BMC Womens Health. 2021 Oct 30;21(1):379. doi: 10.1186/s12905-021-01518-8. PMID 34717608